CLINICAL TRIAL: NCT03528109
Title: Comparison of Patient-Centered Versus Provider-Centered Delivery of Cognitive Behavioral Treatment (CBT) for Pediatric Anxiety and Obsessive Compulsive Disorder (OCD)
Brief Title: Improving Access to Child Anxiety Treatment
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bradley Hospital (Other)
Collaborators: Brown University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHS-2017C1-6400
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety Disorders; Pediatric Disorder; Anxiety; OCD; Phobia; Agoraphobia; Generalized Anxiety; Generalized Anxiety Disorder; Selective Mutism; Separation Anxiety; Social Anxiety; Social Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Phobic Disorders; Agoraphobia; Generalized Anxiety Disorder; Mutism; Anxiety, Separation; Phobia, Social; Panic Disorder | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient-centered home CBT (Experimental): 60 minute office-based exposure therapy with a PhD psychologist once per month and a 90 minute community-based CBT with a mobile exposure coach three times per month for a total of four visits per month (once per week)
  Interventions: Behavioral: Exposure Therapy
- Provider-centered (Active Comparator): 60 minute office-based exposure therapy with a PhD psychologist four times per month (once per week)
  Interventions: Behavioral: Exposure Therapy
- patient-centered telehealth CBT (Experimental): 60 minute telehealth exposure therapy with a PhD psychologist once per month and a 90 minute telehealth CBT with a mobile exposure coach three times per month for a total of four visits per month (once per week). Patient-centered telehealth was closed when the recruitment goal was met in May 2021.
  Interventions: Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy — A type of Cognitive Behavioral Therapy shown to be effective in the treatment of pediatric OCD and anxiety
  Other Names: Exposure-Focused Cognitive Behavioral Therapy (CBT), ExRP

SUMMARY:
There is strong evidence that cognitive behavioral therapy (CBT) with exposure is the preferred treatment for youth with anxiety disorders, but outpatient services that provide this type of treatment are limited. Even for those who do have access to anxiety-specific treatment, a traditional outpatient model of treatment delivery may not be suitable. Among the numerous logistical barriers to treatment access and response is the inability to generalize treatment tools to settings outside of the office. Patient-centered (home-based or telehealth; patient-centered telehealth closed as of 5/1/21) treatment models that target symptoms in the context in which they occur could be more effective, efficient, and accessible for families. The present study aims to compare the efficacy, efficiency, and feasibility of patient centered home-based CBT and patient centered telehealth CBT with a traditional office-based model of care. The question proposed, including proposed outcomes, have been generated and developed by a group of hospital, payer, patient and family stakeholders who will also contribute to the iterative process of protocol revision. The investigators anticipate 379 anxious youth to be randomized to receive outpatient treatment using telehealth (patient-centered telehealth closed as of 5/1/21), home-based services, or treatment as usual using a traditional outpatient model. Results of this study are expected to provide evidence for the efficacy and efficiency of patient-centered treatment, as well as increase treatment access and family engagement in the treatment process.

DETAILED DESCRIPTION:
Anxiety disorders are a significant public health problem that cause suffering for youth and their families, derail normal childhood development, and when left untreated persist into adulthood with high societal costs. Cognitive Behavioral Treatment (CBT) including exposure therapy is the treatment of choice, yet multiple barriers limit access to care. Even for families with access to care, traditional provider-centered (office based) treatment presents challenges and can limit effectiveness for many youth and families. Home- and Community-based exposure therapy is efficacious for patients who previously did not improve with provider-centered services, and input from family stakeholders suggests that treatment in these settings is an optimal match for their needs. Patient-centered models involving home visits and provider teams have consistently demonstrated increased treatment accessibility and engagement. However, there has been no comprehensive comparison of exposure delivered by patient-centered teams using home visits versus by provider-centered office visits alone for childhood anxiety. The absence of comparative effectiveness research (CER) data impedes targeted use of patient centered versus traditional outpatient treatment and would better allocate limited resources, provide the best quality care, and help patients and families make educated decisions about their treatment choices. Telehealth has strong evidence for effectiveness for youth with anxiety and OCD when delivered by a licensed provider, with treatment responder rates ranging from 73-82% (Carpenter, et al., 2018; Comer et al., 2017; Storch et al., 2011). Although traditional telehealth treatments can address barriers associated with in-person treatment, it has yet to be leveraged to increase service capacity. The overall goal of this proposal is to compare two models of service delivery, patient-centered delivery (utilizing novel deployment of personnel both in-home and via telehealth, patient-centered telehealth closed as of 5/1/21) vs. traditional provider-centered delivery, of CBT in youth ages 5-18 receiving exposure therapy for anxiety. A total of 379 children will be treated, with 166 (or 167) children randomly assigned to provider-centered, 166 (or 167) assigned to patient-centered in-home, and 46 assigned to patient-centered telehealth treatment conditions. The patient-centered telehealth condition was added in 2020 in response the COVID-19 global pandemic and closed when the recruitment goal was reached in May 2021. Telehealth treatment models are a necessary health system adaptation in the current health crisis, but also may improve access to care post pandemic. We hope including telehealth as a comparator in our service delivery compared effectiveness trial will be highly informative and relevant for the future mental healthcare landscape.

A trained independent evaluator (IE) blind to condition will measure patient and family treatment engagement, anxiety symptoms/severity, and functional impairment at baseline, during active treatment at weeks 6, 12, 18, and 24, and 3- and 6-month follow-up after acute treatment. The primary aims are to compare the relative effectiveness of patient-centered vs. provider-centered treatment for: 1) improving family treatment engagement/satisfaction, 2) reducing anxiety symptoms, and 3) reducing associated disability (quality of life and functional impairment). Secondary outcomes are to understand moderators of treatment response including: severity of illness, caregiver burden/family accommodation, and barriers to treatment access and to explore group differences in time course of response, durability of treatment gains, provider volume/capacity and efficiency in patient centered versus provider centered treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 5-18 inclusive
* primary or co-primary DSM-V diagnosis of anxiety or OCD
* symptom duration of at least 3 months
* outpatient care needed
* presence of a stable parent, or guardian, who can participate in treatment

Exclusion Criteria:

* other primary or co-primary psychiatric disorder which requires initiation of other active current treatment
* documented mental retardation
* thought disorder or psychotic symptoms
* conduct disorder
* acute suicidality
* concurrent psychotherapy
* chronic medical illness that would preclude their active participation in treatment
* treatment with psychotropic medication that is not stable

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 379 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale | In-treatment and follow-up (6-12 months)
  The CY-BOCS is a measure of obsessive compulsive symptoms and severity. The Obsession Rating Scale measures 5 domains of obsessional severity on a scale from 0 (no impairment) to 4 (extreme impairment.) The Compulsion Rating Scale measures 5 domains of compulsion severity on a scale from 0 (no impairment) to 5 (extreme impairment.) The total range of OCD severity is reported on a scale from 0-40, with a higher score indicating greater severity.
Pediatric Anxiety Rating Scale | In-treatment and follow-up (6-12 months)
  The PARS is a measure of anxiety symptoms and severity. The Anxiety Severity Items are 7 questions meant to assess the frequency of anxiety symptoms and associated impairment. Items are measured on a scale from 0 (none) to 5 (extreme).The total range of anxiety severity is reported on a scale from 0-35, with a higher score indicating greater severity.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire-8 | In-treatment and follow-up (6-12 months)
  The CSQ-8 measures consumer satisfaction with mental health services; satisfaction is measured using 8 items on a scale from 1 (Poor) to 4 (Excellent). Total satisfaction ranges from 8-32, with a high score indicating greater satisfaction.
Clinical Global Impression Scales | In-treatment and follow-up (6-12 months)
  The CGI is a clinician-rated measures of global severity and improvement. The Severity of illness scale reports the severity of current symptoms on a scale from 1 (not at all ill) to 7 (among the most extremely ill patients.) The Global Improvement Scale tracks improvement since treatment initiation on a scale from 1 (very much improved) to 7 (very much worse). The highest possible score on either scale is 7, indicating extreme severity or worse treatment outcome.
Child Sheehan Disability Scale | In-treatment and follow-up (6-12 months)
  The CSDS measures the extent to which anxiety symptoms interfere with functioning. The Disability Scale measures the degree to which anxiety impacts school, social, and home life on a scale from 0 (Not at all) to 10 (very, very much.) Total anxiety-related impairment ranges from 0-30, with higher scores indicating greater impairment.
Homework Compliance Form | Up to 6 months
  The measure tracks both the quality and quantity of homework completed between treatment sessions. This form has been used previously by our research group in large-scale treatment trials, and has been helpful in determining barriers to homework completion.
Exposure Guide | Up to 6 months
  The Exposure Guide is a exposure therapy fidelity/quality tool completed by study therapists. This tool collects information regarding the use of specific therapeutic tools during exposures.
Therapeutic Alliance Scales for Caregivers and Parents (TASCP) | Up to 6 months
  The TASCP is a 12-item measure of therapeutic alliance between a caregiver and his/her child's therapist. This measure assesses the bond and collaboration between caregiver and therapist. Each item is rated using a scale from 0: "not true" to 4: "very much true."
Therapeutic Alliance Scales for Children-Revised (TASC-r) | Up to 6 months
  75 The TASC-r is a 12-item measure of therapeutic alliance between a child and his/her therapist. This measure assesses the degree of affective bond between child and therapist, as well as amount of therapeutic task collaboration. Each item is rated using a scale from 0: "not true" to 4: "very much true."
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) | In-treatment and follow-up (6-12 months)
  The PQ-LES-Q is a 13-item measure of child functioning in life that uses a 5-point ratings scale, with higher scores indicating better quality of life. This measure has both parent and child versions, assessing the same items from both child and parent perspectives. The measure assesses quality of the child's life in a variety of domains.
Top Problems Assessment (TPA) | In-treatment and follow-up (6-12 months)
  The TPA is designed to independently solicit from youth and parent the top 3 problems they feel are most important to address in treatment. This is an idiographic measure of impairment that is driven by the individual needs and desires of the consumer. Respondents rate how much each problem bothers them from 0 ("not at all") to 10 (very, very much).
Caregiver Strain Questionnaire (CSQ) | In-treatment and follow-up (6-12 months)
  The CSQ assesses parent perceptions of the extent to which caring for a child with emotional problems affects several domains, including family life and relationships, demands on time, financial strain, disruption of social life, worry, guilt, and fatigue. This is a 21-item self-report measure that calls for parents to rate the extent of strain for each item using a 0 ("not at all") to 4 ("very much") scale.
Barriers to Treatment Questionnaire - Parent Version (BTQ-P) | In-treatment and follow-up (6-12 months)
  The BTQ-P is a 28-item measure adapted from the BTQ to assess parent perceptions of barriers to accessing treatment for their child's anxiety. The measure is completed at the outset of treatment and assesses such domains as logistic and financial barriers, stigma, and aspects of treatment. Items are rated on a 0 ("not at all true") to 2 ("mostly true") scale.
Pediatric Accommodation Scale-Parent Report (PAS-PR) | In-treatment and follow-up (6-12 months)
  The PAS-PR is a 5-item questionnaire assessing the frequency and interference associated with accommodating the child's anxiety. Each item is followed by a series of common examples to illustrate the principle of accommodation for parents. Responses for frequency include 0 (never), 1 (rarely), 2 (occasionally), 3 (often), and 4 (always). Response options for interference due to accommodation include 0 (none), 1 (mild), 2 (moderate), 3 (severe), and 4 (extreme).
Randomization Debrief | Administered at baseline
  We will record reactions from caregivers and child to treatment assignment using this clinician-rated measure. It includes capturing both verbatim responses from caregivers and child, as well as asking for interviewer impressions reactions from caregivers and child to treatment group assignment following randomization. The clinician also records the likelihood that the family will remain in the study and adhere to study protocols.
Treatment Expectancy | Administered at baseline
  This measure is a 3-item self-report questionnaire that captures parental beliefs about the efficacy about each treatment condition (office-based or home/community-based) using a scale from 1:"I expect my child will be very much improved," to 7: "I expect my child will be very much worse." The parent is also asked to select which treatment option would be best for their family. There is also a patient version of this measure used to capture patient beliefs about the efficacy about each treatment condition (office-based or home/community-based) using the same scale. The patient is asked to select which treatment option they believe would be best for them and their family. The patient version of this measure will be completed by youth 12+.
The Social Responsiveness Scale, Second Edition (SRS-2) | Administered at baseline and at discharge (up to 6-months)
  The SRS-2 is a 65-item self-report measure administered to caregivers or teachers to assess their perception of the presence of a child's social impairment. This measure is used to evaluate children aged 4-18 years old. Items are rated on a scale from 1 ("not true") to 4 ("almost always true").
Affective Reactivity Index - Parent Version (ARI-P) | In-treatment and follow-up (6-12 months)
  The ARI-P is a 7-item parent report questionnaire assessing child's irritability. The items are each given a rating of: "not true," "somewhat true" or "certainly true".
Affective Reactivity Index - Self Report (ARI-S) | In-treatment and follow-up (6-12 months)
  The ARI-S is a 7-item self-report report questionnaire assessing irritability. The items are each given a rating of: "not true," "somewhat true" or "certainly true".
Distress Intolerance Index | In-treatment and follow-up (6-12 months)
  The Distress Intolerance Index is a 10-item self-report report questionnaire assessing the inability to tolerate negative somatic and emotional states. Items are rated on a 5-point scale from "very little" (0) to "very much".
Parent Accommodation Scale (PAS) | In-treatment and follow-up (6-12 months)
  The PAS is a 12-item questionnaire assessing the frequency of and beliefs about parental accommodation. The frequency of parental accommodation is measured on a scale from "Never/Almost Never" (0), to "Always/Almost Always" (3). The beliefs about parental accommodation are measured on a scale from "Strongly Disagree" (0), to "Strongly Agree" (3).
Feedback Forms - Caregiver and Child Versions | Administered only at discharge, up to 6-months into study
  The feedback form is a 3-item self-report questionnaire that asks caregivers or child which treatment group their family was in and for open-ended feedback about their experience in the study (i.e. what did they really like, what would they change, general suggestions/ comments). All responses on this survey are received anonymously. Caregivers and children complete separate feedback forms. Children 8+ will complete the child version of this measure.
End of Treatment Form | Administered only at discharge, up to 6-months into study
  This form captures whether the patient ended treatment before or at 6 months, as well as the reasons for discontinuation (e.g., scheduling, transportation, financial, treatment fit, symptoms) that apply. This form also gathers information about whether referrals were provided to the family upon study discharge.
Sharing Study Findings | Administered only at discharge, up to 6-months into study
  This 7-item measure asks for participants' caregivers to discuss to whom they would like the findings of the study to be disseminated (i.e., local policy makers, educators, etc.). Additionally, it asks for information on how they would like findings to be shared (i.e., via social media, presentations, etc.) as well as caregivers to share highlights of their experience in the study.
Treatment Attendance | Up to 6 months
  We will record the rate of session reschedules, cancellations and no-shows, along with the overall number of sessions attended. We will also document the reason why a scheduled appointment does not occur using the Treatment Cancellation Form.
Reasons for Treatment Discontinuation form | Administered only at discharge, up to 6-months into study
  This is a case record form that documents any change in patient status (e.g., drop-out and premature termination) and the reasons for such changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Freeman, PhD, Principal Investigator — Warren Alpert Medical School of Brown University
Locations (1):
- Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No